CLINICAL TRIAL: NCT06426108
Title: Association of Low-intensity Laser and a Remineralizing Agent in Controlling the Pain of Incisor Molar Hypomineralization in Children: a Randomized, Placebo-controlled, Triple-blind Clinical Trial
Brief Title: Interventions to Control Hypersensitivity Pain in Teeth With Insisive Molar Hypomineralization
Acronym: LBIARHMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Lucas Masaru Marubayashi, Clinical Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 63035222.3.0000.5419; FORP-USP (Other: UNIVERSITY OF SAO PAULO RIBEIRÃO PRETO FACULTY OF DENTISTRY)
Record Dates: First submitted 2024-05-12; First posted 2024-05-23 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Molar Incisor Hypomineralization
Keywords: Molar Incisor Hypomineralization; low-intensity Laser; Dental hypersensitivity
MeSH Terms: conditions — Molar Hypomineralization | interventions — Fluorides, Topical

STUDY DESIGN:
Intervention Model Description: Randomized placebo controlled triple blind clinical trial
Who Masked: Outcomes Assessor
Masking Description: Triple blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Low-Intensity Laser 1J + Fluoride Varnish (Active Comparator): The tooth will undergo low-intensity laser irradiation in continuous mode, employing a wavelength of 808 nm, a power output of 100 mW, a dose of 1 Joule, and a fluence of 35 J/cm^2. The laser will be positioned perpendicular to the tooth surface, targeting the cervical third of the vestibular surface (both mesial and distal aspects), as well as the center of the lesion, with an activation time of 1 Joule (equivalent to 10 seconds). In conjunction with the laser therapy, a fluoride varnish (Duraphat®, containing 22,600 ppm F, manufactured by Colgate) will be utilized as an adjuvant. Application will be facilitated using a microbrush, ensuring coverage over the entire extent of the lesion for 30 seconds. Following the interventions, patients will be advised to refrain from consuming hard foods and to postpone tooth brushing for at least four hours post-application of the varnish, adhering to the manufacturer's guidelines.
  Interventions: Drug: Fluoride Varnishes; Radiation: Low-Intensity Laser 1J
- Low-Intensity Laser 1J + Placebo (Placebo Comparator): The tooth will be subjected to low-intensity laser irradiation in continuous mode, employing a wavelength of 808 nm, a power output of 100 mW, a dose of 1 Joule, and a fluence of 35 J/cm^2. The laser will be positioned perpendicular to the tooth surface, targeting the cervical third of the vestibular surface (both mesial and distal aspects), as well as the center of the lesion, with an activation time of 1 Joule (equivalent to 10 seconds). As an adjunct to the laser therapy, a placebo varnish, devoid of the active ingredient (fluoride), will be utilized. The varnish will be applied with the assistance of a microbrush, ensuring coverage over the entire length of the lesion for 30 seconds. Following the interventions, patients will be advised to abstain from consuming hard foods and to postpone tooth brushing for at least four hours post-application of the varnish.
  Interventions: Drug: Varnishes placebo; Radiation: Low-Intensity Laser 1J
- Low-Intensity Laser 2J + Fluoride Varnish (Experimental): The tooth will undergo low-intensity laser irradiation in continuous mode, utilizing a wavelength of 808 nm, a power output of 100 mW, a dose of 2 Joules, and a fluence of 35 J/cm^2. The laser will be positioned perpendicularly in contact with the tooth surface, targeting the cervical third of the vestibular surface (both mesial and distal aspects), as well as the center of the lesion, with an activation time of 2 Joules (equivalent to 20 seconds). As an adjunct to the laser therapy, a fluoride varnish (Duraphat®, containing 22,600 ppm F, manufactured by Colgate) will be utilized. The varnish application will be facilitated using a microbrush, ensuring coverage over the entire length of the lesion for 30 seconds. Following the interventions, patients will be instructed to refrain from consuming hard foods and to postpone tooth brushing for at least four hours after applying the varnish, in accordance with the manufacturer's recommendations.
  Interventions: Drug: Fluoride Varnishes; Radiation: Low-Intensity Laser 2J
- Low-Intensity Laser 2J + Placebo. (Sham Comparator): The tooth will undergo low-intensity laser irradiation in continuous mode, employing a wavelength of 808 nm, a power output of 100 mW, a dose of 2 Joules, and a fluence of 35 J/cm^2. The laser will be positioned perpendicular to the tooth surface, targeting the third cervical region of the vestibular surface (both mesial and distal aspects), as well as the center of the lesion, with an activation time of 2 Joules (equivalent to 20 seconds). As an adjunct to the laser therapy, a placebo varnish, devoid of the active ingredient (fluoride), will be utilized.The varnish will be applied with the assistance of a microbrush, ensuring coverage over the entire length of the lesion for 30 seconds. Following the interventions, patients will be advised to abstain from consuming hard foods and to postpone tooth brushing for at least four hours post-application of the varnish.
  Interventions: Drug: Varnishes placebo; Radiation: Low-Intensity Laser 2J

INTERVENTIONS:
Drug: Fluoride Varnishes — the investigators will utilize a fluoride varnish with a concentration of 22,600 ppm F. The application will be facilitated using a microbrush, ensuring thorough coverage over the entire length of the lesion for a duration of 30 seconds. Following application, the varnish will be finished with water to create a film on the tooth surface. After completing the interventions, patients will receive instructions to refrain from consuming hard foods and to postpone tooth brushing for at least four hours, adhering to the manufacturer's recommendations.
  Arms: Low-Intensity Laser 1J + Fluoride Varnish; Low-Intensity Laser 2J + Fluoride Varnish
Drug: Varnishes placebo — the investigators will apply a placebo varnish without the active ingredient (fluoride), ensuring that it is packaged identically to the fluoride varnish and has the same taste and texture, thus maintaining consistency in application. The varnish will be applied using a microbrush, spreading it evenly over the entire length of the lesion for a duration of 30 seconds. Following the interventions, patients will receive instructions to avoid consuming hard foods and to delay tooth brushing for at least four hours after applying the varnish.
  Arms: Low-Intensity Laser 1J + Placebo; Low-Intensity Laser 2J + Placebo.
Radiation: Low-Intensity Laser 1J — The tooth will undergo low-intensity laser irradiation in continuous mode, employing a wavelength of 808 nm, a power output of 100 mW, a dose of 1 Joule, and a fluence of 35 J/cm^2. The laser will be positioned perpendicular to the tooth surface, targeting the cervical third of the buccal surface (both mesial and distal aspects), as well as the center of the lesion.
  Arms: Low-Intensity Laser 1J + Fluoride Varnish; Low-Intensity Laser 1J + Placebo
Radiation: Low-Intensity Laser 2J — The tooth will undergo low-intensity laser irradiation in continuous mode, employing a wavelength of 808 nm, a power output of 100 mW, a dose of 2 Joules, and a fluence of 35 J/cm^2. The laser will be positioned perpendicular to the tooth surface, targeting the cervical third of the buccal surface (both mesial and distal aspects), as well as the center of the lesion.
  Arms: Low-Intensity Laser 2J + Fluoride Varnish; Low-Intensity Laser 2J + Placebo.

SUMMARY:
Molar incisor hypomineralization (MIH) manifests as a qualitative, demarcated defect in tooth enamel of systemic origin, predominantly affecting one or more permanent first molars, and potentially extending to the incisors. One significant challenge in managing this enamel anomaly is hypersensitivity, leading to discomfort and pain in affected patients. Low-intensity laser therapy, alone or combined with other modalities, appears promising in alleviating pain associated with MIH. This study aims to assess the efficacy of low-intensity laser therapy using varied parameters, in conjunction with a remineralizing agent, for pain management in children with molar incisor hypomineralization. Participants aged 6 to 12 years will be recruited, with a total of 88 teeth diagnosed with MIH, presenting a sensitivity score ≤3 on the Visual Analog Scale (VAS) and a score ≤1 on the Schiff Cold Air Sensitivity Scale (SCASS). The teeth will be randomly assigned to one of four groups (n=22 each): Group I (GI): L-1J + VF, Group II (GII): L-1J + VP, Group III (GIII): L-2J + VF, and Group IV (GIV): L-2J + VP. Here, 'L' denotes low-intensity laser application at different parameters (1J and 2J), combined with either fluoride varnish (VF) or a placebo varnish (VP). Interventions and assessments will be conducted initially, after 48 hours, and at 1 and 2 weeks post-treatment. Patients will undergo re-evaluation at 2, 4, 8, and 12 weeks following interventions. Statistical analyses will be performed with a 95% confidence level (α = 0.05).

DETAILED DESCRIPTION:
A randomized clinical trial will be carried out involving children aged 6 to 12 years, with a total of 88 teeth diagnosed with MIH, presenting a sensitivity score ≤3 on the visual analogue scale (VAS) and a score ≤1 on the Schiff Cold Air Sensitivity Scale (SCASS). ). Inclusion criteria will require the presence of at least one erupted permanent molar with an occlusal surface free of gingival tissue, demonstrating IMH with sensitivity. Additionally, participants must provide informed consent forms signed by parents or guardians, along with consent forms signed by children. Exclusion criteria include decayed teeth, atypical carious lesions, teeth that have other enamel defects such as fluorosis, enamel hypoplasia, amelogenesis imperfecta or enamel malformations associated with syndromes, ongoing orthodontic treatment, cognitive disorders in patients, desensitizing treatments recent use in the last 3 months, previous use of anti-inflammatory and/or analgesic medications, teeth diagnosed with MIH presenting post-eruptive dentin fractures, atypical restorations, atypical caries, sensitivity scores >3 on the visual analogue scale (VAS) and scores > 1 on the Schiff Cold Air Sensitivity Scale (SCASS).

For the diagnosis of MIH, the investigators will employ the criteria outlined by the European Academy of Pediatric Dentistry, which includes assessment of demarcated opacities, post-eruptive enamel defects, atypical restorations, teeth lost due to MIH, and incompletely erupted teeth. The sample size was determined based on the anticipated outcome of pain reduction following treatment, with an expected 60% reduction. Calculation was conducted with a confidence level of 95% and a power of 80%.

Following the application of the inclusion and exclusion criteria, each group will consist of a total of 88 teeth, randomly assigned to one of four groups: GI, GII, GIII, and GIV. The interventions for each group will be as follows:

GI: Low-Intensity Laser 1J (10 seconds) + Fluoride Varnish. GII: Low-Intensity Laser 1J (10 seconds) + Placebo. GIII: Low-Intensity Laser 2J (20 seconds) + Fluoride Varnish. GIV: Low-Intensity Laser 2J (20 seconds) + Placebo.

To administer laser therapy, the investigators will utilize a low-intensity infrared diode laser (Therapy EC, DMC Equipamentos Ltda., São Carlos, Brazil) operating in continuous mode, emitting at a wavelength of 808 nm with a power output of 100 mW. The dosage will be set at either 1 or 2 Joules, with a fluence of 35 J/cm^2. Both the operator and the patient will wear personal protective equipment (PPE) during the procedure. The tooth will be irradiated perpendicular to the tooth surface, targeting the cervical third of the buccal surface (both mesial and distal aspects), as well as the center of the lesion. Activation time will be either 10 or 20 seconds, corresponding to 1 or 2 Joules respectively, depending on the assigned group. To ensure consistency, even if the laser is activated for 1 Joule (equivalent to 10 seconds), the laser tip will be maintained in place for a standardized duration of 20 seconds, the maximum activation time, as confirmed by a stopwatch in all applications to ensure reliability.

As an adjunct to LBI, the investigators will use a fluoride varnish (FV) and a placebo varnish (PV) without the active ingredient, ensuring that they are in identical packaging with the same taste and texture. Both will maintain the same method of application. The FV used will be Duraphat® (22,600 ppm F, Colgate). The application of both FV and PV will be conducted according to each respective group. Application will be facilitated using a microbrush, spreading it over the entire lesion area for 30 seconds. After the interventions, patients will be instructed not to consume hard foods and to refrain from brushing their teeth for at least four hours following varnish application, adhering to the manufacturer's recommendations.

Following all tests, the data will undergo normality analysis (Shapiro-Wilk test) and homoscedasticity assessment (Levene's test) to determine the suitability of parametric statistics. Therefore, for all variables, one-way ANOVA will be employed, followed by Tukey's post-hoc test for group comparisons. Demographic data will be evaluated using Pearson's chi-square test. Friedman's test may be utilized for multiple comparisons (sensitivity assessments), and the Wilcoxon test for paired comparisons. Analyses will be conducted using the statistical software SPSS 12.0 (SPSS Inc., Chicago, IL, USA). All tests will be performed at a 95% confidence level (α = 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 12 years old
* Teeth diagnosed with MIH, exhibiting at least one erupted permanent molar with the occlusal surface devoid of gingival tissue and showing sensitivity associated with MIH with sensitivity score ≤3 on the Visual Analogue Scale (VAS) and score ≤1 on the Self-Consensus Assessment scale symptoms and signs (SCASS).
* Children who have the cognitive ability to answer the tests.
* Children who obtained authorization from their parents or guardians, through a signed free and informed consent form.

Exclusion Criteria:

* Decayed or restored teeth.
* Teeth with other enamel defects, such as fluorosis, enamel hypoplasia, amelogenesis imperfecta or enamel malformations associated with syndromes, as well as those undergoing orthodontic treatment.
* Patients with cognitive impairments that prevent responsiveness to the test.
* Children who have undergone desensitizing treatment in the last 3 months.
* Children who use anti-inflammatory and/or analgesic medications before starting treatment.
* Teeth that have a sensitivity score >3 on the visual analogue scale (VAS) and a score >1 on the Schiff Cold Air Sensitivity Scale (SCASS).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Gradual change of hypersensitivity on the visual analogue scale. | Gradual reduction after 48 hours, and at 1 and 2 weeks post-treatment and remaining stable during follow-ups of 2, 4, 8, and 12 weeks following interventions
  Applying the low intensity laser of 1 joule (10 seconds) in infrared light in continuous mode, using a wavelength of 808 nm, power of 100 mW, dose of 1 or 2 Joules and fluence of 35 J/cm2. As an adjuvant to fluoride varnish (22,600 ppm F), we expect an improvement in hypersensitivity assessed by the visual analogue scale, ranging from 0 (no pain) to 10 (worst possible pain), so that applications performed after 48 hours will decrease, and in 1 and 2 weeks post-treatment, remaining stable during follow-ups at 2, 4, 8 and 12 weeks after interventions. This expectation arises from the known mechanisms of laser action in controlling inflammation and providing analgesia. Furthermore, we also anticipate that fluoride varnish will exert its remineralizing effects, contributing to the overall treatment of the disease.

SECONDARY OUTCOMES:
Gradual change of hypersensitivity on the Schiff Cold Air Sensitivity Scale | Gradual reduction after 48 hours, and at 1 and 2 weeks post-treatment and remaining stable during follow-ups of 2, 4, 8, and 12 weeks following interventions
  Applying the low intensity laser of 1 joule (10 seconds) in infrared light in continuous mode, using a wavelength of 808 nm, power of 100 mW, dose of 1 or 2 Joules and fluence of 35 J/cm2. As an adjuvant to fluoride varnish (22,600 ppm F), we expect improvement in hypersensitivity assessed by the Schiff Cold Air Sensitivity Scale, ranging from 0 (the child does not respond to the stimulus) to 3 (the child responds to the stimulus, moves away and requests immediate suspension of the stimulation), so that it decreases with applications carried out after 48 hours, and at 1 and 2 weeks post-treatment, remaining stable during follow-ups at 2, 4, 8 and 12 weeks after the interventions. This expectation arises from the known mechanisms of laser action in controlling inflammation and providing analgesia. Furthermore, we also anticipate that fluoride varnish will exert its remineralizing effects, contributing to the overall treatment of the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucas Masaru Marubayashi, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Muniz RSC, Carvalho CN, Aranha ACC, Dias FMCS, Ferreira MC. Efficacy of low-level laser therapy associated with fluoride therapy for the desensitisation of molar-incisor hypomineralisation: Randomised clinical trial. Int J Paediatr Dent. 2020 May;30(3):323-333. doi: 10.1111/ipd.12602. Epub 2019 Dec 23. PMID 31808584
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31808584/

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT06426108/SAP_000.pdf